CLINICAL TRIAL: NCT04468152
Title: Increased Dietary Intake and Serum Levels of Advanced Glycation End Products Are Associated With Diabetic Macular Edema
Brief Title: Advanced Glycation End Products Are Associated With Diabetic Macular Edema
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Sedat Arslan, Principal Investigator, Hacettepe University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Screening
Other Study IDs: GO 18/562
Record Dates: First submitted 2020-07-03; First posted 2020-07-13 (Actual); Last update posted 2020-07-13 (Actual); Status verified 2020-07

CONDITIONS: Diabetic Macular Edema; Diabetes Mellitus, Type 2
Keywords: advanced glycation end products; diabetic macular edema; nutrition
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Case (Experimental)
  Interventions: Behavioral: Dietary habits and intake
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Dietary habits and intake — Optical coherence tomography (OCT) withdrawals and central foveal thickness (CFT) evaluations of those included in the study were made by the doctor and directed to the dietician (researcher). The dietary intake of participants was assessed using a validated quantitative food frequency questionnaire (QFFQ) (21). The total food intake was then converted to total nutrient intake based on the food's nutrient profile. Standardized food recipes for Turkey and the Nutrition Information System (BEBIS) program, which is a food composition database for nutrient estimation, were used to determine the average daily energy and nutrient intake for each participant.
  Arms: Case

SUMMARY:
Diabetic macular edema can develop at all stages of diabetic retinopathy, causing visual impairment and blindness. Modern diets are high in advanced glycation end products (dAGEs), derived from processing methods, exerting a pivotal role in promoting diabetic retinopathy risk. In this cross-sectional study, we investigate the relationship between dietary and serum levels of AGEs and DME in type 2 diabetic subjects.

DETAILED DESCRIPTION:
This was a cross-sectional study was carried out in the Hacettepe University Hospital, Department of Ophthalmology, between July 2018 and February 2019.

While benefiting from the results of the previous studies, the sample size of the research was type 1 error level α = 0.05 and type 2 level β = 0.20. The power analysis was statistically calculated using NCCS PAS 11 program. The present study was conducted with 90 patients: 50 case-patients (DM with DME) and 40 control patients (DM without DME). Excluded from the study were those under the age of 18 years, with no diagnosis of Type 2 DM, without any anti-diabetic agent, with any disease other than DME and DR that may affect the retina, with any disease that may affect the retina for the control group, with corneal, lens or vitreous opacification preventing Optical coherence tomography (OCT) withdrawal, with any systemic disease other than DM and hypertension, with a history of eye surgery, and with blindness or infection in the eye, along with those recently diagnosed with diabetes (<1 year) and those with special diets.

This the study was conducted in accordance with the Declaration of Helsinki Ethical Principles.

OCT withdrawals and CFT evaluations of those included in the study were made by the doctor and directed to the dietician (researcher). Demographic data and the dietary habits were collected through standardized face-to-face interviewer-assisted questionnaires. The bodyweight and height of patients were measured using a calibrated body composition analyser and weight scales by researcher. BMI was evaluated based on the WHO classification. Waist and hip circumference was also measured and evaluated in terms of high risk of developing chronic diseases. Hypothesis: If the waist/hip ratio is ≥0.85 for women and ≥0.90 for men, the risk of developing chronic diseases increases.

Diabetic macular edema (DME) Examination After a detailed systemic and ophthalmological history was taken from all subjects by the doctor, the best-corrected visual acuity level was measured using an ETDRS chart. A fundus examination was performed with a 90 D lens after anterior segment examination and pupil dilation with a biomicroscope. A spectral-domain OCT (Spectralis OCT, Heidelberg Engineering, Heidelberg, Germany) was applied for the evaluation of CFT. After a minimum of eight hours of fasting, approximately 5 ml of peripheral venous blood was collected from the antecubital region in the HÜTF Ophthalmology Clinic between 08:00 and 10:00.

Assessment of dietary intake and dietary AGEs The dietary intake of participants was assessed using a validated quantitative food frequency questionnaire (QFFQ) (including about 110 food items take 20-25 minutes to complete). Foods were classified into eight categories: dairy products, meat products, fruits, vegetables, bread and cereals, beverages, and desserts. Also, questions were asked to patients about traditional cooking methods to calculate dietary AGE intakes. Such as what cooking methods do they cook the foods? How long do they cook the food? Standardized food recipes for Turkey and the Nutrition Information System (BEBIS) program were used to calculate the average daily energy and nutrient intake for each participant. Meanwhile, to assess dietary AGEs from the QFFQ, each food's contribution to dAGEs intake was calculated based on the Advance Glycation End Products in Foods Table published by the Uribarri et al., which comprises data on 549 food items.

Sample Collection and Analysis The serum samples collected during the research were delivered to the laboratory while preserving the cold chain. The enzyme-labeled immune "Enzyme-Linked Immunosorbent Assay (ELISA)" test was performed with biologists of the company using a Biotek 800TS device. While analyzing the samples, Human CML Elisa Kit 96 tests for serum AGE and Human RAGE Elisa Kit 96 test kits for serum RAGE were used. Carboxymethyl lysine (CML) was considered as the AGE parameter, being the most easily detected and the most abundant type of AGE in humans. The minimum detectable dose of CML in humans is typically less than 15.6 pg/ml.

ELIGIBILITY:
Inclusion Criteria:

* Included from the study were those over the age of 18 years, with diagnosis of Type 2 DM.

Exclusion Criteria:

* Excluded from the study were those under the age of 18 years, with no diagnosis of Type 2 DM, without any anti-diabetic agent, with any disease other than DME and DR that may affect the retina, with any disease that may affect the retina for the control group, with corneal, lens or vitreous opacification preventing Optical coherence tomography (OCT) withdrawal, with any systemic disease other than DM and hypertension, with a history of eye surgery, and with blindness or infection in the eye, along with those recently diagnosed with diabetes (<1 year) and those with special diets.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2018-07-07 (Actual); Primary Completion 2019-01-10 (Actual); Study Completion 2019-01-10 (Actual)

PRIMARY OUTCOMES:
We hypothesize that the AGEs levels of the DME group would found be higher than in the control group. | 3 months
  The serum samples collected during the research were delivered to the laboratory while preserving the cold chain. The enzyme-labelled immune "Enzyme-Linked Immunosorbent Assay (ELISA)" test was performed with biologists of the company using a Biotek 800TS device. While analyzing the samples, Human CML Elisa Kit 96 tests for serum AGE is used. Carboxymethyl lysine (CML) was considered as the AGE parameter, being the most easily detected and the most abundant type of AGE in humans. The minimum detectable dose of CML in humans is typically less than 15.6 pg/ml.
We hypothesize that the dietary intake of AGEs wolud be higher in the DME group. | 1 month
  The dietary intake of participants was assessed using a validated quantitative food frequency questionnaire (QFFQ). The total food intake was then converted to total nutrient intake based on the food's nutrient profile. Standardized food recipes for Turkey and the Nutrition Information System (BEBIS) program, which is a food composition database for nutrient estimation, were used to determine the average daily energy and nutrient intake for each participant. These values were subsequently compared with the recommended daily allowance values to determine the status of meeting energy and nutrient requirements. After that, the percentages meeting the requirements were calculated. Meanwhile, to assess dietary AGEs from the QFFQ, each food's contribution to dAGEs intake was calculated based on the Advance Glycation End Products in Foods Table published by the Uribarri et al.
We hypothesize that neck circumference correlated significantly with DME. | 1 month
  The neck circumference of the participants will be measured by the researcher Sedat Arslan with a calibrated tape measure on a centimeter scale.

SECONDARY OUTCOMES:
We hypothesize that the sRAGE levels were higher in the DME group. | 3 months
  The serum samples collected during the research were delivered to the laboratory while preserving the cold chain. The enzyme-labelled immune "Enzyme-Linked Immunosorbent Assay (ELISA)" test was performed with biologists of the company using a Biotek 800TS device. While analyzing the samples,Human RAGE Elisa Kit 96 test kits for serum RAGE were used.

CONTACTS AND LOCATIONS:
Overall Officials: Sibel Kadayıfçılar, Prof.Dr., Study Chair — Hacettepe University; Gülhan Samur, Prof.Dr., Study Director — Hacettepe University; Dila Kırağı, Dr., Study Chair — Hacettepe University
Locations (1):
- Hacettepe University Hospital Department of Ophthalmology Polyclinic, Ankara, Altındağ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No